CLINICAL TRIAL: NCT01778075
Title: A Single Dose, Open-Label, Randomized, Two-Way Crossover Pivotal Study to Assess the Bioequivalence of a New ULTRACET ER Tablet With Respect to a Marketed ULTRACET ER Tablet Under Fasted Condition
Brief Title: A Study to Assess the Bioequivalence of a New ULTRACET Extended Release (ER) Tablet With Respect to a Marketed ULTRACET ER Tablet Under Fasted Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100924; TRAMCTPAI1003 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Healthy; Ultracet extended release (ER); Tramadol hydrochloride; Acetaminophen; Bioequivalence
MeSH Terms: interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence AB (Experimental): Treatment A: Newly developed Ultracet ER; Treatment B: Marketed Ultracet ER
  Interventions: Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Newly developed ULTRACET ER); Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Marketed ULTRACET ER)
- Treatment sequence BA (Experimental): Treatment A: Newly developed Ultracet ER; Treatment B: Marketed Ultracet ER
  Interventions: Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Newly developed ULTRACET ER); Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Marketed ULTRACET ER)

INTERVENTIONS:
Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Newly developed ULTRACET ER) — Single oral dose of newly developed ULTRACET ER, (Tramadol HCl/Acetaminophen 75/650 mg), administered under fasted condition.
Drug: Tramadol HCl 75 mg/Acetaminophen 650 mg (Marketed ULTRACET ER) — Single oral dose of marketed ULTRACET ER, (Tramadol HCl/Acetaminophen 75/650 mg), administered under fasted condition.

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a newly developed ULTRACET extended-release (ER) tablet of tramadol hydrochloride and acetaminophen, to the current marketed ULTRACET ER tablet, in healthy participants under fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate
* Must agree to use an adequate contraception method as deemed appropriate by the investigator (e.g., vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Body mass index (weight [kg]/height2 [m]2) between 18.5 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Blood pressure (after the participant is sitting for 5 minutes) between 90 and 140 mm Hg systolic, inclusive, and no higher than 90 mm Hg diastolic
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac function, including sinus rhythm, pulse rate between 45 and 90 bpm, QTc interval <= 450 ms, QRS interval of <110 ms, PR interval <200 ms, and morphology consistent with healthy cardiac function

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic (blood) disease, coagulation disorders (including any abnormal bleeding), lipid abnormalities, significant lung disease (including bronchospastic respiratory disease), diabetes mellitus, kidney or liver insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening (or at admission to the study center) as deemed appropriate by the investigator
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for oral contraceptives and hormonal replacement therapy within 14 days before the first dose of the study drug is scheduled
* History of, or reason to believe a participant has a history of, drug or alcohol abuse within the past 5 years

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of racemic tramadol (Period 1) | Up to 48 hours following the administration of study drug on Day 1 of Period 1
Plasma concentrations of acetaminophen (Period 1) | Up to 48 hours following the administration of study drug on Day 1 of Period 1
Plasma concentrations of racemic tradamdol (Period 2) | Up to 48 hours following the administration of study drug on Day 1 of Period 2
Plasma concentrations of acetaminophen (Period 2) | Up to 48 hours following the administration of study drug on Day 1 of Period 2

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | Approximately 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: A Single-Dose, Open-Label, Randomized, Two-Way Crossover Pivotal Study to Assess the Bioequivalence of a New ULTRACET ER Tablet With Respect to a Marketed ULTRACET ER Tablet Under Fasted Conditions — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3592&filename=CR100924_CSR.pdf